CLINICAL TRIAL: NCT05596240
Title: The Effects of Dry Needling on Muscle Blood Flow of the Infraspinatus in Individuals with Shoulder Pain - a Randomized Controlled Trial
Brief Title: Dry Needling and Shoulder Muscle Blood Flow, Motions, and Pain Sensitivity in Individuals with Shoulder Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Jace Brown, Principal Investigator, Texas Woman's University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-FY2022-438
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dry Needling; Shoulder Pain
Keywords: dry needling; shoulder pain; pain pressure threshold
MeSH Terms: conditions — Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Pre-test Post-Test Design
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not be told whether they are assigned to the interventional or sham group. The outcomes (blood flow, pain pressure threshold, and range of motion) will be assessed by an investigator blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry Needling (Experimental): Individuals with shoulder pain will receive dry needling to the two to four most tender points in the infraspinatus based on examiner palpation
  Interventions: Other: Dry Needling
- Sham Dry Needling (Placebo Comparator): Individuals with shoulder pain will receive sham dry needling to two points in the muscle belly of the infraspinatus near the insertion and below the midpoint of the spine of the scapula
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry Needling — A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the MTrP of the infraspinatus muscles. Once the needle has been inserted, the technique described by Hong (1994) will be used. The needle will be pistoned in an up and down motion within the infraspinatus muscle at approximately 1Hz for 10 seconds with the aim of eliciting local twitch responses.
  Arms: Dry Needling
Other: Sham Dry Needling — Streitberger Placebo-needles (Asia-med, Las Vegas, NV) will be used to perform the intervention for participants in the sham DN group. These needles have been reported to be indistinguishable from real needles. The device consists of a plastic tube with a blunted tip needle that allows for the sensation of a prick without penetrating the skin. The sham needle produces a sensation, which causes the participant to feel as if the needle enters the skin, while maintaining similar patient-therapist contact time and total intervention time.
  Arms: Sham Dry Needling

SUMMARY:
Shoulder pain is one of the most common reasons people consult with their primary health care provider, and 40-50% of these patients with shoulder pain continued to complain of persistent symptoms after 6 to 12 months. It has been suggested that the presence of myofascial trigger points (MTrPs) may contribute to the chronicity of shoulder symptoms. An MTrP is a hyperirritable taut band of tissue within a muscle that produces pain when stimulated MTrPs are common in patients with shoulder disorders and occur most often in the infraspinatus muscle of a painful shoulder MTrPs were associated with an acidic biochemical environment with elevated levels of inflammatory mediators, neuropeptides, and proinflammatory cytokines such as bradykinin and calcitonin g-related peptide. It was hypothesized that metabolic demands on muscle and capillary constrictions may contribute to the development of MTrPs. To date, only a few studies have examined the vascular environment of MTrPs and surrounding areas before and after dry needling. No studies have yet examined whether dry needling would change blood flow in patients with shoulder pathology. Therefore, the purpose of this pilot study is to examine the effect of dry needling on blood flow of the infraspinatus muscle using color Doppler imaging in individuals with shoulder pain. The secondary purpose is to examine the effect of DN on shoulder motion and sensitivity to pressure in individuals with shoulder pain.

DETAILED DESCRIPTION:
RESEARCH DESIGN This pilot study will be a single-blinded randomized comparison trial with two groups: (1) the group that will receive real DN, and (2) a placebo group that will receive sham DN. The research design will be a prospective two-way (2 x 2) mixed design to examine the effects of DN on blood flow (i.e., peak systolic velocity, end diastolic velocity, resistive index, pulsatile index) of the infraspinatus, shoulder range of motionss of internal rotation and external rotation, and PPTs of the infraspinatus. The two independent variables are: (1) group with two levels (DN and sham DN groups), and (2) time with two levels (baseline and immediately after the intervention) for the peak systolic velocity, end diastolic velocity, resistive index, pulsatile index of the infraspinatus, shoulder internal rotation, shoulder external rotation, and PPTS of the infraspinatus.

INSTRUMENTATION A color-Doppler ultrasonographic scanner and a curvilinear transducer (Sonosite Edge; Sonosite, Inc., Bothell, WA) will be used to measure blood flow of the infraspinatus muscle. The curvilinear probe (5-2MHz) has ability to capture images up to 30 cm in depth. A standard goniometer with 1° increments will be used to measure shoulder ROMs. Standard goniometric measurements have shown good-to-excellent reliability for shoulder internal and external ROMs.23 A hand-held computerized pressure algometer (Medoc ltd., Ramat Yishai, Israel) will be used to measure the PPT over the infraspinatus muscle. The algometer consists of a 1 cm2 round-tip that will be pressed perpendicular to the skin of the infraspinatus muscle at a rate of 40kPa/s until the first perception of pain or discomfort detected by the participant. The participant will be able to stop the test with a press of a button upon feeling the first sensation of pain or discomfort. This device has shown to have high test-retest reliability (intraclass correlation coefficients = 0.70-0.94) in the shoulder and neck muscles.

PROCEDURE At the beginning of the visit, all participants will be asked for demographic information and their pain-related characteristics, including location, duration, intensity at onset, and intensity currently, at best, and at worst in the previous 24-hours using the NPRS. After the subjective information is gathered, an investigator will assess for the presence of MTrP based on palpation. The participant will be placed in the prone position with arms resting at their side. The examiner will palpate the infraspinatus muscle belly for the presence of a taut band, a hypersensitive spot, and reproduction of the participants symptoms.11 Al-Shenqiti and Oldham25 demonstrated high reliability (k=0.86) with palpation for the presence or absence of the taut band, spot tenderness, and/or referred pain sensation.

Once the participant is determined eligible, they will be asked to complete the Quick Disability of Arm Shoulder Hand (QuickDASH) questionnaire to determine their self-reported disability and function (Appendix C).26 Next, the three outcome measures will be collected, including blood flow parameters, shoulder ROMs, and PPTs. If the participant has bilateral shoulder pain, the most painful shoulder will be tested. If both shoulders are equally painful, a coin-flip will be used to determine the side on which testing will be performed. The outcome measurements will be administered in an order of shoulder ROMs, followed by PPT and blood flow parameters before the DN intervention. Following the intervention, the outcome measurements will be collected in a reverse order of blood flow parameters, PPT, and shoulder ROM to minimize the position changes and to capture immediate changes of blood flow. These outcomes will be assessed by an investigator blinded to the intervention assignment.

SHOULDER RANGE OF MOTION ROM testing will be performed while the participant is lying supine with the shoulder at 90° abduction and 10° of horizontal abduction and elbow at 90°flexion. The examiner will be responsible for all the measurements. The center of rotation of the goniometer will be placed over the olecranon while one arm of the goniometer will be positioned along the length of the ulna, aligned with the ulnar styloid process. The other arm will be positioned perpendicular to the ground. For both measurement of internal and external rotation, scapular compensation will be monitored by using the thumb on the coracoid process and fingers along the spine of the scapula. Each measurement will be repeated three times with the average measurements used for data analysis.

PRESSURE PAIN THRESHOLD MEASUREMENT During the PPT testing, the participant will be placed in the prone position with upper extremities relaxed at their sides. PPT of the infraspinatus muscle will be tested in the muscle belly 1.5 inches below the midpoint of the spine of scapula. The participants will be given a stop button and will be instructed to stop the test as soon as the pressure becomes uncomfortable or painful, and not to allow a painful or uncomfortable sensation to continue. The participants will be familiarized with the algometer, which will consist of a single trial on the non-painful side to ensure that the participant understands the process. A total of three trials will be performed and the average of three trials will be used for data analysis. The PPT of the infraspinatus muscle has been shown to have good-to-excellent intraday, interday, intrarater, and interrater reliability.27,28

ULTRASOUND IMAGING Each participant will remain in the same position for ultrasound imaging. The ultrasound transducer will be placed perpendicular to the infraspinous fossa to visualize arterioles or arteries in the vicinity of the MTrPs and to quantify the velocity of flow at the MTrPs of the infraspinatus. The location of the transducer will be outlined after initial placement to ensure consistent placement of the transducer between trials as well as before and after DN. The spectral Doppler waveforms will be analyzed to trace the velocities throughout the cardiac cycle. The peak systolic (PSV), end diastolic velocity (EDV), resistive index (RI), and pulsatile index (PI) will be calculated using software available on the device. On a Doppler waveform, the PSV corresponds to each "peak" within the spectral window, whereas the EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak. These values will be used to calculate the RI with the formula RI = (PSV - EDV)/PSV and the PI with the formula PI = (PSV EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle. A reliability study is currently underway to establish the test-retest reliability of this ultrasound testing protocol (TWU IRB # IRB-FY2022-349).

INTERVENTION Following the baseline testing, the participants will be randomly assigned to either the real DN group or sham DN group. A large opaque envelope containing 40 cards, 20 cards marked "DN" and 20 marked "sham DN" will be used for random assignment. Each participant will be randomly assigned based on the card drawn from the envelope. The group assignment will be performed by the treating physical therapist. If a participant withdraws from the study, a card for the group to which they are assigned will be returned to the envelope.

For the real DN group, the technique described by Hong14 will be used to needle the two to four MTrPs in the infraspinatus muscle based on the results of the examiner's palpation. A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the MTrP of the infraspinatus muscles. Once the needle has been inserted, the needle will be pistoned in an up-and-down motion within the infraspinatus muscle at approximately 1Hz for 10 seconds with the aim of eliciting local twitch responses.

Streitberger Placebo-needles (Asia-med, Las Vegas, NV) will be used to perform the intervention for participants in the sham DN group. These needles have been reported to be indistinguishable from real needles. The device consists of a plastic tube with a blunted tip needle that allows for the sensation of a prick without penetrating the skin. The sham needle produces a sensation, which causes the participant to feel as if the needle enters the skin, while maintaining similar patient-therapist contact time and total intervention time.29

REASSESSMENT Immediately following the intervention, the three outcomes will be collected from all participants in the following order to minimize position changes: blood flow parameters, PPT, and shoulder ROMs. Additionally, any adverse events, such as bruising, nausea, dizziness, or post-needling soreness following the dry needling procedures will be assessed immediately. If bleeding occurs, the participant will be informed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 with unilateral nonspecific shoulder pain based on participants' self-reported pain level of greater than or equal to 2/10 on the Numeric Pain Rating Scale (NPRS) in last 24 hours
* non-traumatic origin of pain
* presence of at least one MTrP with referral pain pattern in the infraspinatus muscle determined through palpation.

Exclusion Criteria:

* systemic joint disease (e.g. rheumatoid arthritis)
* evidence of red flags (e.g. signs of current fracture or history of fracture to scapula, glenoid or proximal humerus, infection, tumor, incontinence, or paresthesias)
* cancer
* neurological disorders
* neuropathy
* Raynaud's disease
* pregnancy
* previous shoulder surgery
* repeated infection (e.g. systemic infection, red skin, fever, individuals who are visibly unwell or toxic in appearance)
* immunocompromised disease (e.g., diabetes mellitus, HIV, AIDS, lupus)
* inability to maintain the testing and treatment positions (i.e., supine and prone-lying) for 15 minutes at a time.
* bleeding disorders (e.g. hemophilia)
* use of anti-coagulants (e.g. vitamin K antagonists, direct oral anticoagulants, and low molecular weight heparins)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Peak Systolic Velocity | Change from baseline PSV immediately
  On a Doppler waveform, the PSV corresponds to each "peak" within the spectral window. These values will be used to calculate the RI with the formula RI = (PSV - EDV)/PSV.
Resistive Index (RI) | Change from baseline RI immediately
  Resistive Index is used to assess the resistance in a pulsatile vascular system.The RI is defined by the the formula RI = (PSV - EDV)/PSV.
Pulsatile Index (PI) | Change from baseline PI immediately
  Pulsatility index (PI) is defined as the difference between the peak systolic flow and minimum diastolic flow velocity, divided by the mean velocity recorded throughout the cardiac cycle. It is a non-invasive method of assessing vascular resistance with the use of Doppler ultrasonography. PI is defined with the formula PI = (PSV - EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle.
End Diastolic Velocity (EDV) | Change from baseline EDV immediately
  EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak.

SECONDARY OUTCOMES:
Pain Pressure Thresholds (PPT) | Change from baseline PPT immediately
  Pressure pain threshold (kPa) is a quantitative sensory test, used to measure deep muscular tissue sensitivity to mechanical pressure stimuli. The test determines the amount of pressure over the infraspinatus in which a steadily increasing non-painful pressure stimulus turns into a painful pressure sensation.
Shoulder Range of Motion | Change from baseline shoulder range of motion immediately
  shoulder range of motion of internal and external rotation is the number of degrees of motion measured using standard goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jace A Brown, DPT, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University T. Boone Pickens Institute of Health Sciences - Dallas Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the summary data are published. Data obtained through this study may be provided to qualified researchers with academic interest in Dry Needling. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Bron C, Dommerholt J, Stegenga B, Wensing M, Oostendorp RA. High prevalence of shoulder girdle muscles with myofascial trigger points in patients with shoulder pain. BMC Musculoskelet Disord. 2011 Jun 28;12:139. doi: 10.1186/1471-2474-12-139. PMID 21711512
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Diaz-Rodriguez L, Gonzalez-Iglesias J, Palacios-Cena D, Arroyo-Morales M. Changes in pain and pressure pain sensitivity after manual treatment of active trigger points in patients with unilateral shoulder impingement: a case series. J Bodyw Mov Ther. 2011 Oct;15(4):399-404. doi: 10.1016/j.jbmt.2010.12.003. Epub 2011 Jan 17. PMID 21943613
- [Background] Ge HY, Fernandez-de-Las-Penas C, Yue SW. Myofascial trigger points: spontaneous electrical activity and its consequences for pain induction and propagation. Chin Med. 2011 Mar 25;6:13. doi: 10.1186/1749-8546-6-13. PMID 21439050
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Sandberg M, Lundeberg T, Lindberg LG, Gerdle B. Effects of acupuncture on skin and muscle blood flow in healthy subjects. Eur J Appl Physiol. 2003 Sep;90(1-2):114-9. doi: 10.1007/s00421-003-0825-3. Epub 2003 Jun 24. PMID 12827364
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Nascimento JDSD, Alburquerque-Sendin F, Vigolvino LP, Oliveira WF, Sousa CO. Absolute and Relative Reliability of Pressure Pain Threshold Assessments in the Shoulder Muscles of Participants With and Without Unilateral Subacromial Impingement Syndrome. J Manipulative Physiol Ther. 2020 Jan;43(1):57-67. doi: 10.1016/j.jmpt.2019.04.002. Epub 2020 Feb 13. PMID 32061418